CLINICAL TRIAL: NCT04871802
Title: A Prospective, Randomized, Comparative Study in Two Groups to Assess the Effect of the Use of a Dietary Supplement Taxifolin Aqua on the Recovery Period After COVID Pneumonia and on the Biological Age
Brief Title: Effect of the Dietary Supplement Taxifolin Aqua on the Recovery Period After COVID-19 Pneumonia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Pirogov Russian National Research Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: COVID-AQUA-1
Record Dates: First submitted 2021-03-21; First posted 2021-05-04 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-03

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Taxifolin Aqua group (Experimental): Taxifolin Aqua 30 mg per day in addition to standard therapy
  Interventions: Dietary Supplement: Taxifolin Aqua
- Control group (No Intervention): No intervention

INTERVENTIONS:
Dietary Supplement: Taxifolin Aqua — Dietary supplement
  Arms: Taxifolin Aqua group

SUMMARY:
Objective of the study is to evaluate the effect of Taxifolin Aqua therapy on the indicators of respiratory function, the state of the arterial wall, the contractile function of the myocardium, as well as to assess the effect of Taxifolin Aqua therapy on markers of biological age, quality of patients life.

DETAILED DESCRIPTION:
The study will include 100 patients who had covid pneumonia 3 months ago. If the inclusion / exclusion criteria are met, the patient is asked to sign an informed consent to participate in the study. Consenting patients are randomized to an intervention group or a control group. The control group (n = 50) will receive standard therapy, patients from the intervention group (n = 50) will be prescribed Taxifolin Aqua 30 mg per day in addition to standard therapy. Patients will be randomized to the control and main group using random number spreadsheets, assuming that the control and main groups will be homogeneous in the main demographic and clinical parameters. Patient monitoring will be carried out within 2 months from the date of inclusion. A follow-up visit is scheduled in 2 months. During the study, the patient will be regularly monitored for tolerance and safety of therapy with Taxifolin Aqua.

ELIGIBILITY:
Inclusion Criteria:

Patients of both sexes who had covid pneumonia 3 months ago and signed an informed consent and aged 18+.

Exclusion Criteria:

Standard contraindications to Taxifolin Aqua use.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-05-10 (Estimated); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Dynamics of spirometry indices | In 2 months after recruitment
  spirometry
Dynamics of ECHO CG | In 2 months after recruitment
  ECHO CG
Dynamics of pulse wave velocity | In 2 months after recruitment
  applanation tonometry
Dynamics of augmentation index | In 2 months after recruitment
  applanation tonometry

SECONDARY OUTCOMES:
Dynamics of biological age | In 2 months after recruitment
  Laboratory indicators

CONTACTS AND LOCATIONS:
Overall Officials: Irina Strazhesko, MD, PhD, Principal Investigator — Clinical Reserach Center for Gerontology
Locations (1):
- Russian Clinical Research Center for Gerontology, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No